CLINICAL TRIAL: NCT00388713
Title: Radiation Induced Atherosclerosis in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: ASBCO5- HMO-CTIL
Record Dates: First submitted 2006-10-15; First posted 2006-10-17 (Estimated); Last update posted 2007-05-16 (Estimated); Status verified 2005-12

CONDITIONS: Abnormalities, Radiation-Induced; Atherosclerosis; Breast Cancer
Keywords: Radiation therapy; Radiation-Induced Atherosclerosis; Carotid Artery Diseases; Breast Cancer; Intima Media thickening Ultrasound
MeSH Terms: conditions — Abnormalities, Radiation-Induced; Atherosclerosis; Breast Neoplasms; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: carotid intima-media thickening ultrasound

SUMMARY:
Radiation induced accelerated atherosclerosis is a well known entity that occurs in different regions, according to the therapy delivered.It is usually begins to be clinically evident several years after the radiation incident, as there is sufficient functional reserve to these vessels.Our proposal is aimed to better characterize this side effect. For that purpose, we have chosen to study women who received radiation to the breast, in which part of the carotid in the irradiated side was in the high energy radiation field. We will use Intima Media Thickening ultrasound to study the pattern of atherosclerosis plaque formation in radiated carotid arteries as compared to non-irradiated carotid arteries in women who are receiving radiation therapy for breast cancer.

DETAILED DESCRIPTION:
Radiation induced atherosclerosis in Breast Cancer patients

Radiation induced accelerated atherosclerosis is a well known entity that occurs in different regions, according to the therapy delivered. This process takes a couple of years to develop. Therefore, the most affected populations are the long term survivors of potentially curative cancers such as Hodgkins lymphoma 1, 2, head and neck cancers 3-6, pelvic cancers (both prostate cancer and cervical cancer) 7, and breast cancer8-14. The mechanism of damage is thought to be direct endothelial damage, which is most significant about 6 months post XRT, followed by inflammation, cholesterol plaque formation and intimal thickening. This cascade, as well as the pathological findings, are similar to what is seen in natively occurring AS. However, in the post XRT setup, it is not limited to one part of the artery and usually encompasses the entire circumference of the radiated segment15-17.

The accelerated atherosclerosis resulting from radiation usually begins to be clinically evident several years after the radiation incident, as there is sufficient functional reserve to these vessels. However, changes can be seen much sooner, and some studies have shown significant changes as soon as one year after the initial insult 2, 18.

Literature reports suggest as high as 77.5% of symptomatic carotid stenosis (on risky regions of common carotid and internal carotid arteries) as compared to 21.6% on the matched control group (consisting of newly diagnosed patients with similar risk factors)18. A retrospective review from Philadelphia on 413 treated patients found RR for stroke of 2, as compared with the general population (matched for risk factors) from the Stockholm database5. Data from the Netherlands suggested risk for stroke as high as 5 times as compared to the matched group without cancer. The analysis was done on patients who received the treatment before 60 yo (the comparison was not made to the general population as these patient are usually smokers and drinkers and are usually at a higher risk to begin with, however XRT increases this already high risk by 5).

A new emerging technique of Carotid Intima-Media Thickening (IMT) has demonstrated the impact of radiation (2.2 Vs 0.7mm in controls)6.

Our proposal is aimed to better characterize this side effect. For that purpose, we have chosen to study women who received radiation to the breast, in which part of the carotid in the irradiated side was in the high energy radiation field. The contralateral artery, which received only trace of scattered radiation, can serve as the internal control. This is not the case in head and neck patients, who usually receive a high dose of radiation to both sides of the neck. The number of early breast cancer patients who received adjuvant radiation is relatively high, a factor which may help us reach the accrual goal much faster. Subsequently we are planning to proceed in a consecutive study and to try to pharmacologically interfere with progression of the AS, and perhaps even prevent it.

Intima Media Thickening US is a non-invasive US technique that is available at Hadassah University Medical Center and will be performed in this study in order to detect the degree of AS in affected and non affected arteries.

The suggested study will consist of two populations. Group 1 are women who received radiation for breast cancer in the past at various time intervals and the Group 2 are women with newly diagnosed breast cancer.

Markers and biochemistry tests that might elucidate predisposing and contributing factors for developing AS will also be done and analyzed on all patients. The latter could be a target for treatment and a surrogate to the treatment efficacy, side effects, and cancer progression (i.e. cholesterol levels, hypertension, hypothyroidism, etc.)

ELIGIBILITY:
Inclusion Criteria:

* women 18-85 Y.O.
* received or about to receive unilateral breast and supraclavicular radiation therapy
* No evidence of disease

Exclusion Criteria:

* prisoners

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2006-10; Study Completion 2010-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amichay Meirovitz, MD, Principal Investigator — Hadassah University Hospital, Jerusalem, Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Adams MJ, Hardenbergh PH, Constine LS, Lipshultz SE. Radiation-associated cardiovascular disease. Crit Rev Oncol Hematol. 2003 Jan;45(1):55-75. doi: 10.1016/s1040-8428(01)00227-x. PMID 12482572
- [Background] Cheng SW, Ting AC, Lam LK, Wei WI. Carotid stenosis after radiotherapy for nasopharyngeal carcinoma. Arch Otolaryngol Head Neck Surg. 2000 Apr;126(4):517-21. doi: 10.1001/archotol.126.4.517. PMID 10772307
- [Background] Dorresteijn LD, Kappelle AC, Boogerd W, Klokman WJ, Balm AJ, Keus RB, van Leeuwen FE, Bartelink H. Increased risk of ischemic stroke after radiotherapy on the neck in patients younger than 60 years. J Clin Oncol. 2002 Jan 1;20(1):282-8. doi: 10.1200/JCO.2002.20.1.282. PMID 11773180